CLINICAL TRIAL: NCT06304883
Title: Long-term Extension of a Phase 3, Multicenter, Randomized, Double-Blind, Placebo- Controlled Study of the Efficacy, Safety, and Biomarker Effects of ALZ-801 in Subjects With Early Alzheimer's Disease and APOE4/4 Genotype
Brief Title: Long-term Extension of Phase 3 Study of ALZ- 801 in APOE4/4 Early AD Subjects
Acronym: APOLLOE4-LTE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alzheon Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALZ-801-AD351
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Early Alzheimer's Disease
Keywords: Dementia; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease; Dementia; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: This is a multi-center, open-label, single group, long-term extension study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: ALZ-801 (Experimental): ALZ-801 265 mg BID tablet orally. Subjects will take one 265 mg tablet of ALZ-801 in the evening during the first 4 weeks of the study; thereafter, they will take one 265 mg tablet BID.
  Interventions: Drug: Experimental: ALZ-801

INTERVENTIONS:
Drug: Experimental: ALZ-801 — ALZ-801 265 mg BID tablet orally.

SUMMARY:
This study is being conducted to evaluate the long-term safety and efficacy of ALZ-801 in Early Alzheimer's disease (AD) subjects with the APOE4/4 genotype. This is an open-label trial of treatment with ALZ-801.

DETAILED DESCRIPTION:
This is a long-term extension study of the Phase 3, multicenter, randomized, double-blind, placebo-controlled study of the efficacy, safety, and imaging biomarker effects of ALZ-801 in subjects with Early Alzheimer's Disease and APOE4/4 genotype. Subjects who at initial screening for the Phase 3 study were 50-80 years old, had a clinical diagnosis of AD, carried the APOE4/4 genotype, and were at the early stage of disease (Early AD], who complete at least 78 weeks of the Phase 3 study while on study medication, were eligible for enrollment. Subjects will be treated for 104 weeks with ALZ-801, followed by a 4-week safety follow-up visit after the last dose of ALZ-801. Clinical trial sites, subjects and their study partner will remain blinded to the treatment (ALZ-801 or placebo) that they received in the core Phase 3 study. The primary efficacy outcome assessment is a measure of cognition (ADAS-Cog 13). Additional measures of global and functional impairments will also be assessed. Imaging and biomarkers of AD and neurodegeneration will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed the Week 78 of the Phase 3 core study (ALZ-801-AD301) while on study drug.
* Subject has a reliable study partner who has sufficient contact with the subject to be able to provide accurate information about the subject's cognitive and functional abilities.

Exclusion Criteria:

* Significant worsening of medical conditions that may preclude completion of this study.
* Evidence of symptomatic or new moderate-severe radiologic ARIA at baseline.
* Has received (or plans to receive) amyloid antibodies since completing Phase 3 core study (ALZ-801-AD301).
* Subject taking any prohibited medications per protocol.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Primary cognitive efficacy endpoint 1 | Week 104
  Change from baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale 13 (ADAS-Cog 13), from baseline of Phase 3 core study (ALZ-801-AD301) to Week 52 and Week 104 of this long-term extension study (ALZ-801-AD351).
Primary cognitive efficacy endpoint 2 | Week 104
  Change from baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale 13 (ADAS-Cog 13), from baseline of this study to Week 52 and Week 104.
Incidence, Nature, and Severity of Treatment Emergent Adverse events (TEAEs) | Week 104
  Safety and tolerability as measured by incidence, nature and severity of treatment emergent adverse events (TEAE), serious TEAE, and TEAE leading to withdrawal.
Primary imaging biomarker endpoint 1 | Week 104
  Change from baseline in total hippocampal volume (mm3) as measured by Magnetic Resonance Imaging (MRI), from baseline of the Phase 3 core study (ALZ-801-AD301) to Week 52 and Week 104 of this long-term extension study (ALZ-801-AD351).
Primary imaging biomarker endpoint 2 | Week 104
  Change from baseline in total hippocampal volume (mm3) as measured by Magnetic Resonance Imaging (MRI), from baseline of this study to Week 52 and Week 104.

SECONDARY OUTCOMES:
Secondary functional efficacy endpoint | Week 104
  Change from baseline of the Phase 3 core study, and from baseline and from Week 52 of this study, in Disability Assessment for Dementia scores.
Secondary functional efficacy endpoint | Week 104
  Change from baseline of the Phase 3 core study, and from baseline and from Week 52 of this study, in Amsterdam - Instrumental Activities of Daily Living scores.
Secondary global assessment efficacy endpoint | Week 104
  Change from baseline of the Phase 3 core study, and from baseline and from Week 52 of this study, in Clinical Dementia Rating - Sum of Boxes (CDR-SB) scores.
Secondary cognitive efficacy endpoint 1 | Week 104
  Change from baseline of the Phase 3 core study, and from baseline and from Week 52 of this study, in Alzheimer's Disease Assessment Scale - Cognitive Subscale 11.
Secondary cognitive efficacy endpoint 2 | Week 104
  Change from baseline of the Phase 3 core study, and from baseline and from Week 52 of this study, in Neuropsychiatric Inventory.
Secondary cognitive efficacy endpoint 3 | Week 104
  Change from baseline of the Phase 3 core study, and from baseline and from Week 52 of this study, in Mini-Mental State Examination.
Secondary imaging biomarker endpoint | Week 104
  Change from baseline of the Phase 3 core study (ALZ-801-AD301) and from baseline of this long-term extension study (ALZ-801-AD351) in cortical thickness, whole brain volume and ventricular volume (mm3) as measured by Magnetic Resonance Imaging (MRI) to Weeks 26, 52, 78 and 104.
Secondary fluid biomarker endpoint | Week 104
  Change from baseline of the Phase 3 core study, and from baseline and from Week 52 of this study in plasma p-tau181, Aβ 42, Aβ 40, GFAP, and NfL levels.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Abushakra, MD, Principal Investigator — Alzheon Inc.
Locations (41):
- United States (29):
  - Xenoscience, Inc., Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - ATP Clinical Research, Costa Mesa, California
  - Torrance Clinical Research Institute, Lomita, California
  - Sutter Health, Sacramento, California
  - JEM Research Institute, Headlands Site, Atlantis, Florida
  - K2 Medical Research, LLC, Maitland, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Charter Research, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - ALZ Research and Treatment Center (A.R.T.C.), Stuart, Florida
  - ALZ Research and Treatment Center (A.R.T.C.), Wellington, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Columbus Memory Center, Columbus, Georgia
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Headlands Research Eastern MA, Plymouth, Massachusetts
  - Advanced Memory Research Center, Toms River, New Jersey
  - Neurological Associates of Albany, Albany, New York
  - NYU Alzheimer's Disease Research Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Triad Clinical Trials, Greensboro, North Carolina
  - AMC Research, Matthews, North Carolina
  - Center for Cognitive Health, Portland, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - UT Health Science Center at Houston, Houston, Texas
  - Re:Cognition Health, Fairfax, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- Canada (5):
  - OCT Research ULC (dba Okanagan Clinical Trials), Kelowna, British Columbia
  - Centricity Research, Halifax, Nova Scotia
  - Recherches Neuro-Hippocampe Inc., d/b/a Ottawa Memory Clinic, Ottawa, Ontario
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - Toronto Memory Program, Toronto, Ontario
- United Kingdom (7):
  - Re-Cognition Health Ltd Plymouth, Plymouth, Devon
  - Re-Cognition Health Ltd London, London, Greater London
  - NeuroClin Glasgow Ltd, Motherwell, North Lanarkshire
  - Re-Cognition Health Ltd Guildford, Guildford, Surrey
  - Re-Cognition Health Ltd Birmingham, Birmingham, West Midlands
  - Re-Cognition Health Ltd Bristol, Bristol
  - Re-Cognition Health Ltd Winchester, Winchester